CLINICAL TRIAL: NCT00149136
Title: Evaluation of Imatinib (GLIVEC) After Induction Therapy in Patients Aged More Than 55 Years With Philadelphia Positive Acute Lymphoblastic Leukaemia (Ph+ ALL) : a Non Randomised, Controlled, Open, Multicentric, International Phase II Clinical Study (CSTI 571 AFR09 Trial)
Brief Title: Treatment of Philadelphia-Positive Acute Lymphocytic Leukemia (Ph+ ALL) in the Elderly With Imatinib Mesylate (STI571) and Chemotherapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2002.280
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Acute Lymphocytic Leukemia,; Ph+,; elderly patients,; Imatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib

SUMMARY:
ALL patients aged 55 years or older were treated with steroids during one week and Ph+ve cases were then offered a specific therapy including an induction treatment with steroids, cyclophosphamide, daunorubicin and vincristine, followed, irrespective of response to induction chemotherapy, by imatinib, 600 mg daily, combined with intermittent steroids during 2 months. Patients in complete response (CR) were then given 10 blocks of alternating chemotherapy, including 2 additional two-month blocks of imatinib, for a total treatment duration of 2 years. Therapy of occult central nervous system leukemia included 5 intrathecal injections of methotrexate and cranial irradiation.

Duration of therapy : 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ph+ ALL patients
* 55 years or older
* Signed written informed consent

Exclusion Criteria:

* CML in transformation
* Concomitant malignancy
* Previous treatment by Imatinib
* Severe organ condition

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-08

PRIMARY OUTCOMES:
Impact of Imatinib on survival in elderly patients with Ph+ALL

SECONDARY OUTCOMES:
Tolerance of Imatinib
Complete remission rate
Minimal Residual Disease after Imatinib treatment
Leukemia free survival
Impact of steroids given before starting chemotherapy
Study of potential resistance mechanisums to Imatinib

CONTACTS AND LOCATIONS:
Overall Officials: Xavier THOMAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Xavier THOMAS, Lyon, France